CLINICAL TRIAL: NCT05451680
Title: A Randomized Study on the Effect of Negative-pressure Wound Therapy on Below-the-knee Skin Cancer Graft Reconstruction Complications
Brief Title: Negative-pressure Wound Therapy on Full-thickness Skin Grafts of the Lower Leg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kirsi Isoherranen, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1020DE009
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Skin Tumor
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: controlled study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative-pressure treatment (Experimental): A negative pressure wound dressing is placed over the skin graft. Patients are started on compression therapy after surgery, unless there are contraindications, and standard oral and written postoperative immobilization and other treatment instructions are given.
  Interventions: Device: Negative pressure device
- Conventional treatment (Active Comparator): A conventional antimicrobial wound dressing is placed on top of the graft. Patients are started on compression therapy after surgery, unless there are contraindications, and standard oral and written postoperative immobilization and other treatment instructions are given.
  Interventions: Procedure: Conventional care

INTERVENTIONS:
Device: Negative pressure device — Negative-pressure therapy postoperatively on the full-thickness skin graft
  Arms: Negative-pressure treatment
Procedure: Conventional care — Conventional dressing postoperatively on the full-thickness skin graft
  Arms: Conventional treatment

SUMMARY:
This randomized controlled non-sponsored trial on 60 patients evaluates if a portable negative-pressure device improves graft-take and decrease the risk of surgical complications for skin-cancer surgeries below the knee.

DETAILED DESCRIPTION:
Annually, 12 000 skin cancers are diagnosed in Finland. This randomized controlled non-sponsored trial evaluate if a portable negative-pressure device improves graft-take and decrease the risk of surgical complications. 60 patients over 18 years of age are included and randomly assigned to either the negative pressure-treatment group or the conventional treatment group. At the control appointment one-week postsurgery, graft take is documented as a primary outcome and any complications (necrosis, infection, hematoma/seroma) and adverse events (pain, skin reactions) as secondary outcomes. Adverse events are evaluated by a phone call 3 weeks postsurgery and based on medical records 3 months postsurgery.

ELIGIBILITY:
Inclusion Criteria:

* from referrals received by the Unit, or from patients undergoing follow-up who have skin cancer (basal cell carcinoma, squamous cell carcinoma or melanoma) or suspected skin cancer below the knee

Exclusion Criteria:

* Toe lesion, bleeding disorder, severe dementia, critical peripheralischemia, or skin disease that is expected to impair wound healing, such as pyoderma gangrenosum

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Graft take | 3 months
  good, partial or poor graft take (%)

SECONDARY OUTCOMES:
Adverse events | 3 months
  Necrosis, infection, hematoma/seroma (%)

CONTACTS AND LOCATIONS:
Locations (1):
- HUS Iho- ja allergiasairaala, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No